CLINICAL TRIAL: NCT01576510
Title: Brain Circuitry and Psychosocial Predictors of PTSD
Brief Title: fMRI Predictors of Treatment Response in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Harvard University (Other); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of Clinical Psyhcology, Research Foundation for Mental Hygiene, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2R01MH072833-04A2 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure (PE) treatment. (Experimental)
  Interventions: Behavioral: Prolonged Exposure (PE)
- Trauma exposed healthy controls (No Intervention): Clinical assessments at baseline, 7 and 10 weeks. fMRI assessments at baseline and 10 weeks.

INTERVENTIONS:
Behavioral: Prolonged Exposure (PE) — Prolonged Exposure (PE) therapy consists of ten 90-minute sessions. Elements of PE include imaginal and in vivo exposure to trauma reminders; breathing retraining; cognitive restructuring; and PTSD psychoeducation. The therapist helps the patient cognitively restructure his/her experience of the traumatic event. Each week the narrative is elaborated, becoming more detailed and exhaustive, until the patient habituates to it, extinguishing the anxiety it formerly aroused.
  Arms: Prolonged Exposure (PE) treatment.

SUMMARY:
To employ a fear learning-extinction paradigm with functional magnetic resonance imaging (fMRI) and skin conductance response (SCR) assessments among patients with posttraumatic stress disorder (PTSD) and trauma exposed healthy controls, aiming to a) clarify neural circuits underlying PTSD and b) to probe brain based predictors of symptomatic improvement in response to Prolonged Exposure (PE) treatment, and first line treatment for PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is highly prevalent and debilitating disorder. It is defined by a fearful response to traumatic events, and its clinical picture includes reexperiencing, arousal, and avoidance to reminders of the exposure. Despite efforts to characterize the pathophysiology of PTSD, no biomarkers have been established that aid in diagnosis, treatment development, or prediction of treatment response.

Several lines of evidence suggest that PTSD symptoms are mediated by dysfunctional processes involving the brain's fear-circuitry network in general, and extinction learning and recall deficits in particular. Based on our preliminary work in applying fear extinction task to healthy humans and patients with PTSD the goal of this renewal RO1 application is to employ an established extinction paradigm with functional magnetic resonance imaging (fMRI) and Skin Conductance Response (SCR) assessments in a large and well characterized sample with PTSD and trauma exposed healthy control (TE-HC) subjects. We plan to clarify circuits underlying PTSD psychopathology and to probe, for the first time, neural circuitry of symptomatic improvement in response to Prolonged Exposure (PE) treatment. This goal is congruent with NIMH strategic plan strategy 1.3 ("identify and integrate biological markers and behavioral indicators associated with mental disorders").

One hundred subjects including 60 individuals with a principal diagnosis of PTSD and 40 trauma exposed healthy controls will be assessed by fMRI and SCR to determine the neural circuitry activation to the fear extinction task. fMRI data will be acquired simultaneously with fear extinction and recall measurement quantified by SCR. All 60 PTSD subjects and 20 randomly assigned TE-HCs subjects will repeat these procedures 10 weeks later, after PTSD subjects have completed 10 weeks of intensive PE treatment. Three months after treatment completion clinical ratings of PTSD severity will be conducted to permit analysis of neural predictors of long term treatment durability.

The aims above will be accomplished through four years of study, conducted by a multi-disciplinary research team, comprised of research scientists from Columbia, Harvard and New York Universities, who have conducted studies in PTSD and structural and functional brain imaging. If successful, the study will produce highly needed information on the neural circuitry which underlies deficient extinction and recall in PTSD, and will provide highly important information about the neural effects of Prolonged Exposure treatment, a first line treatment for PTSD. Together these lines of expected findings will not only advance identification of biomarkers associated with PTSD, but also facilitate identification of biomarkers for clinical reponse to an empirically supported treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 60
2. Current DSM-IV PTSD
3. CAPS score equal or greater than 50.
4. Able to give consent, fluent in English or Spanish.

Exclusion Criteria:

1. History of Axis I psychiatric diagnosis (other than as specified), e.g., psychotic disorder, bipolar disorder, obsessive compulsive disorder (OCD), tic disorder, or eating disorder. Note that comorbid current major depressive disorder will be allowed in up to one half of the PTSD group. This will enable inclusion of this common comorbidity, but also enable an assessment of whether or not the presence of this comorbid diagnosis is driving any observed significant between-group differences.
2. Depression which is antecedent to PTSD; score of > 25 on the Hamilton Rating Scale for Depression (HAM-D-17-item); significant depression and /or depression related impairment that is judged to warrant pharmacotherapy or combined medication and psychotherapy.
3. Individuals at risk for suicide based on history and current mental state.
4. History of substance/alcohol dependence within the past six months, and abuse within past two months
5. Patients who are receiving effective medication for their PTSD and/or depression
6. Antipsychotic, antidepressant, or mood stabilizer medications in the last 4 weeks prior to the study (6 weeks for fluoxetine). Standing daily dosing of benzodiazepine class of medication in the 2 weeks prior to the study (as needed use of benzodiazepines is not an exclusion, but must be clinically judged to tolerate no benzodiazepines for the 72-hour period before each of the fMRI days). Triptan anti-migraine medications. Other medications that may interfere with fear circuitry and fear memory such as blood-brain-barrier-penetrating β-blockers.
7. Pregnancy, or plans to become pregnant during the period of the study.
8. Paramagnetic metallic implants or devices contraindicating magnetic resonance imaging or any other non-removable paramagnetic metal in the body.
9. Formal CBT psychotherapy initiated within 3 months of beginning this study.
10. Medical illness that could interfere with assessment of diagnosis, treatment response or biological measures (SCR, fMRI), including organic brain impairment from stroke, CNS tumor, or demyelinating disease; and renal, thyroid, hematologic or hepatic impairment
11. Current unstable or untreated medical illness, and resting SBP≥140 and DBP≥90 and HR<60 and HR>100
12. Any condition that would exclude clinical MR exam (e.g. pacemaker, paramagnetic metallic prosthesis, surgical clips, shrapnel, necessity for constant medicinal patch, some tattoos)
13. Significant claustrophobia that would preclude ability to remain calm within the MRI scanner

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change over time in Clinician Administered PTSD Scale (CAPS) | Baseline, week 7, week 10, and 3 month follow up
  Structured Interview

SECONDARY OUTCOMES:
Change over time in brain activation patterns as measured by fMRI | Baseline and 10 weeks (post treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Trauma and PTSD Program at New York State psychiatric Institute — http://www.columbiatrauma.org